CLINICAL TRIAL: NCT02880826
Title: Study on the Measurement of Care Safety Culture in French ICU, Correlation With the Characteristics of Morbi-mortality Reviews
Brief Title: Measurement of Care Safety Culture in French ICU, Correlation With the Characteristics of Morbi-mortality Reviews
Acronym: REA-C-SUR
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC13_0028
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Measure the culture of safety in the reanimation units

SUMMARY:
The tools to measure safety culture (CS) have recently become available. No study has focused on the measure in France, apart from pilot studies. intensive services are particularly at risk of serious adverse events occurred (SAEs). Patients who are hospitalized are in fact fragile and precarious clinical condition requires rapid decision taken often. Diagnostic or therapeutic strategies have report "risk-benefit" narrow. They may well be complicated by EIG.Safety of care is a priority in the field of health in general, and especially in intensive care. CS measure in this context seems particularly relevant.

The main objective is to describe the CS intensive care units in France. The study will explore the development of the CS level for the units investigated.

This study will also describe the main features of RMM practiced in intensive care units in France.

ELIGIBILITY:
Inclusion Criteria:

* practicing resuscitation activity (this practice is medical or surgical, pediatric or adult, in public or private sector)
* volunteer to participate in the study (agreement of the head of the unit)
* for which at least 2 matching / references for the study were identified:

  * a medical officer,
  * caregiver responsible (Health Framework).

Exclusion Criteria:

* measurement safety culture done in a period of significant change during a period where the staff and activities of the respondent unit of work is relatively stable.
* the responses of professionals to the questionnaire can be influenced by internal factors in their work unit (recent accident occurred, change of close supervision, personnel changes ...) and by factors external to their unit work (establishment certification period, arrival of a new director, recent media coverage of medical accidents ...).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 60 intensive care units in France. Each unit is estimated that an average of 80 professionals will be subject to the evaluation of the CS (doctors, IDE, assistant nurses, physiotherapists...) and thus nearly 4800 people will be included for the CS measurement.
  Includes: all professionals providing care to patients and working full-time or part-time work in the respondent unit.
Sampling Method: Probability Sample
Enrollment: 4800 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The measure of the CS of intensive care units in France using a validated questionnaire | The planned project duration is 12 months

IPD SHARING:
Plan to Share IPD: Undecided